CLINICAL TRIAL: NCT02357771
Title: Topical Application of Probiotic Lozenge to Reduce Streptococcus Mutans in Plaque Around Orthodontic Brackets
Brief Title: Probiotic Lozenge Reduce Streptococcus Mutans in Plaque in Orthodontic Bracket Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Next Gen Pharma India Pvt. Ltd. (Industry)
Collaborators: Peoples University, Bhanpur, Bhopal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BHO_PERIO-ODB_01
Record Dates: First submitted 2015-02-03; First posted 2015-02-06 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Malocclusion
Keywords: misalignment of the two dental arches; mal-align teeth
MeSH Terms: conditions — Malocclusion | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo Arm (Placebo Comparator): Placebo Lozenges (4 Lozenges per day; 2 lozenges in morning and 2 lozenges in the night). Each placebo lozenge contains all excipients except the active constituent (Lactobacillus brevis CD2)
  Interventions: Drug: Placebo
- Probiotic Arm (Experimental): Lactobacillus brevis CD2 Lozenges (4 Lozenges per day; 2 lozenges in morning and 2 lozenges in the night). Each probiotic lozenge contains not less than 1 billion Colony Forming Unit of L. brevis CD2
  Interventions: Drug: Probiotic (L. brevis CD2 lozenges)

INTERVENTIONS:
Drug: Probiotic (L. brevis CD2 lozenges) — Each Lactobacillus brevis CD2 lozenge contains not less than 1 billion Colony Forming Unit of L. brevis CD2
  Arms: Probiotic Arm
Drug: Placebo — Each placebo lozenge contains all excipients except the active constituent (Lactobacillus brevis CD2)
  Arms: Placebo Arm

SUMMARY:
Advances in orthodontics have improved the quality of appliances and treatment protocols, raising the standard of patient care. However, enamel demineralization is still a problem associated with orthodontic treatment, leading to the formation of white spot lesions; this is a grave concern to orthodontists and patients.

The overall prevalence of white spot lesions among orthodontic patients has been reported to be between 4.9% and 84%.1 When basic oral hygiene is poor, orthodontic appliances create areas of plaque stagnation, especially around brackets, bands, wires, and other attachments. Levels of acidogenic bacteria, present in the plaque, notably Streptococcus mutans (S mutans), are higher in orthodontic patients than in non-orthodontic patients.

This causes demineralization around the brackets and leads to white spot lesions. They are most prevalent around the cervical region of bands in the posterior region, whereas in the anterior region, the lateral incisors in both arches, followed by the canines, are most commonly affected.

ELIGIBILITY:
Inclusion Criteria:

* Orthodontic treatment with the straight wire appliance (MBT, 0.022-in slot; 3M Unitek, Monro- via, Calif).
* Complete permanent dentition (excluding third molars).
* No chewing gum or mouthwash used in the last week and during the study.
* Habit of brushing twice daily with fluoride toothpaste.

Exclusion Criteria:

* Patient with poor periodontal condition.
* Patient with known medical condition e.g. subacute bacterial endocarditis, diabetes, valvular disease, anemia etc.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-04; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Changes in the levels of streptococcus Mutans in the plaque around orthodontic brackets. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Upendra Jain, M. Orth., Study Chair — Peoples College of Dental Sciences & Research Centre, Bhanpur, Bhopal, Madya Pradesh
Locations (1):
- Department of Orthodontics & Dentofacial Orthopaedics, People College Of Dental Sciences & Research Centre, Bhanpur, Bhopal, Madhya Pradesh, India